CLINICAL TRIAL: NCT02289586
Title: Interventional Bronchoscopy Under Noninvasive Ventilation for Central Airway Stenosis
Brief Title: Interventional Bronchoscopy Under Noninvasive Ventilation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Futian People's Hospital (Other)
Collaborators: Science and Technology Innovation Commission of Shenzhen Municipality (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: szkcw-2014-322
Record Dates: First submitted 2014-08-04; First posted 2014-11-13 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-08

CONDITIONS: Noninvasive Positive Pressure Ventilation;; Sedation;; Bronchoscopy；; Interventional；; Central Airway Stenosis
MeSH Terms: interventions — Noninvasive Ventilation; Midazolam; Remifentanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- hypoxemia, central airway stenosis. (Active Comparator): Inclusion Criteria:
  * (a)patients with central airway stenosis need interventional bronchoscopy (b) partial pressure of arterial oxygen (PaO2)/fraction of inspired oxygen (FiO2) ratio less than 300;
  Exclusion Criteria:
  * (a) facial deformity sufficient to preclude mask fitting; (b) upper gastrointestinal bleeding; (c) upper airway obstruction; (d) acute coronary syndromes; (e) tracheostomy or endotracheal intubation(ETI) before admission; (f) need for urgent ETI due to cardiac or respiratory arrest.
  Interventions: Procedure: invasive ventilation; Procedure: interventional bronchoscopy; Drug: general anesthesia(midazolam, fentanyl，rocuronium，propofol and Remifentanil）
- hypoxemia, central airway stenosis (Experimental): Inclusion Criteria:
  * (a)patients with central airway stenosis need interventional bronchoscopy (b) partial pressure of arterial oxygen (PaO2)/fraction of inspired oxygen (FiO2) ratio less than 300;
  Exclusion Criteria:
  * (a) facial deformity sufficient to preclude mask fitting; (b) upper gastrointestinal bleeding; (c) upper airway obstruction; (d) acute coronary syndromes; (e) tracheostomy or endotracheal intubation(ETI) before admission; (f) need for urgent ETI due to cardiac or respiratory arrest.
  Interventions: Procedure: interventional bronchoscopy; Device: noninvasive ventilation; Drug: sedation(dezocine and midazolam)

INTERVENTIONS:
Procedure: invasive ventilation
Procedure: interventional bronchoscopy
Device: noninvasive ventilation
Drug: sedation(dezocine and midazolam)
Drug: general anesthesia(midazolam, fentanyl，rocuronium，propofol and Remifentanil）

SUMMARY:
To evaluate the effect and safety of noninvasive ventilation assisted interventional bronchoscopy for hypoxemia patients with central airway stenosis.

With the sedation and analgesia, noninvasive ventilation assisted interventional bronchoscopy for hypoxemia patients with central airway stenosis is safe and effective, carries high satisfaction rate.

ELIGIBILITY:
Inclusion Criteria:

* (a)patients with central airway stenosis need interventional bronchoscopy. (b) partial pressure of arterial oxygen (PaO2)/fraction of inspired oxygen (FiO2) ratio less than 300;

Exclusion Criteria:

* (a) facial deformity sufficient to preclude mask fitting; (b) upper gastrointestinal bleeding; (c) upper airway obstruction; (d) acute coronary syndromes; (e) tracheostomy or endotracheal intubation(ETI) before admission; (f) need for urgent ETI due to cardiac or respiratory arrest.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-07; Primary Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
The improvement of airway stenosis after the operation | 1 day
The improvement of partial pressure of arterial oxygen (PaO2) after the operation | 1 day

SECONDARY OUTCOMES:
hospitalization expenses | During the period of hospitalization，an expected average of 4 weeks
hypoxemia during the operation | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Futian People's Hospital, Shenzhen, Guangdong, China